CLINICAL TRIAL: NCT03629327
Title: Preventing HIV Infection by Targeting the Immune System Instead of the Virus
Brief Title: Inducing Immune Quiescence the Genital Tract With ASA
Acronym: IIQ-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Keith Fowke, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HS19749(B2016:042); B2016:042 (Other: University of Manitoba)
Record Dates: First submitted 2018-07-30; First posted 2018-08-14 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: HIV
MeSH Terms: interventions — Aspirin; Control Groups

STUDY DESIGN:
Intervention Model Description: Three arms will be followed simultaneously
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ASA 325mg (Active Comparator): Daily uptake of 325mg ASA
  Interventions: Drug: ASA 325mg
- No drug (Active Comparator): no drug
  Interventions: Other: Control Group
- ASA 81mg (Active Comparator): daily uptake of 81mg ASA
  Interventions: Drug: ASA 81mg

INTERVENTIONS:
Drug: ASA 81mg — Participants will be randomized to take 81mg orally on a daily basis for a duration of 6 months
  Other Names: Acetylsalicylic acid 81mg
  Arms: ASA 81mg
Other: Control Group — Participants will be randomized to take nothing on a daily basis for a duration of 6 months
  Other Names: no drug
  Arms: No drug
Drug: ASA 325mg — Participants will be randomized to take 325mg orally on a daily basis for a duration of 6 months
  Other Names: Acetylsalicylic acid 325mg
  Arms: ASA 325mg

SUMMARY:
There are 33.4 million individuals living with HIV/AIDS worldwide. Despite successful HIV prevention strategies such as condom use and reduction of sexual partners, HIV continues to spread at an alarming rate. In 2010, 2.6 millions of new infections were detected. In Sub-Saharan Africa, women represent the two-third of all new infections1. Despite the efforts of the scientific community, there is still no commercial vaccine or microbicide available.

To explain this natural protection against HIV, different mechanisms have been identified. These women have a unique immune phenotype that we called Immune Quiescence. This phenotype is characterized by lower expression of genes involved in cellular activation, lower resting levels of inflammatory cytokine production, lower level of systemic activated T cells, increased levels of systemic T regulatory, increased production of anti-viral anti-protease serpins at the female genital tract and reduced numbers of HIV target cells (mainly CD4+ CCR5+ T cells) in the FGT This project aims to induce an Immune Quiescence phenotype (decreasing immune activation) to prevent HIV infection

DETAILED DESCRIPTION:
HIV is an important global health issue. Globally, HIV is mostly transmitted through heterosexual sexual activity, and women bear the brunt of the pandemic as two-third are in women. New preventive strategies need to be developed to empower women to protect themselves. In Nairobi, Kenya, there are around 27 000 sex workers and despite prevention efforts, HIV incidence is very high in this vulnerable group which serves as catalyzers for HIV transmission to the community. Among those sex workers, despite being at higher risk of infection, some rare individuals remain HIV exposed seronegative (HESN). Over the years, our group has tried to understand this natural protection to HIV infection. The investigators discovered that in HESN individuals, the basal level of activation of the immune system is lower than in other people. This includes having few HIV target cells, mainly CD4+ CCR5+ T cells, in their genital tract. The investigators called this special phenotype Immune Quiescence (IQ). In a recent pilot study (Limiting HIV target cells by Inducing Immune Quiescence in the female genital tract ) the investigators showed that in non-sex worker women it is possible to decrease the proportion of HIV target cells and/or HIV co-receptor at the female genital tract by using anti-inflammatory drugs.

Herein, the investigators are proposing to conduct a follow-up study in female sex workers to determine the best drug formulation and drug size effect on reducing HIV target cell number at the female genital tract (FGT). Participants will receive acetylsalicylic acid (ASA) (81mg/day), ASA (325mg/day), or nothing for five months. At visit 1, the baseline immune activation level of the participants will be determined. In this way, every woman will serve as her own control thereby reducing the variation between tested and control groups. Participants will be randomized and ask to take the drug daily. Participants will be followed on a monthly basis. At each study visit, blood, cervico-vaginal lavage and cervical cells will be taken to determine the level of immune activation. This study is a critical "second step" in the rational development of HIV preventive biomedical method.

ELIGIBILITY:
Inclusion Criteria:

* Age greater of 18 years and less than 45
* Be active in sex work for five years or less
* Uterus and cervix present
* Willing to take daily the study drug (acetylsalicylic acid)
* Willing to undergo pelvic exams
* In general good health, no chronic infection and not taking any anti-inflammatory or immunosuppressors
* Being HIV negative
* Without any cardiovascular disease

Exclusion Criteria:

* Age less than 18 or more than 45
* Breastfeeding
* Pregnant in the last 12 months
* Presence of sexual transmissible disease or bacterial vaginosis at enrollment
* Menopausal
* Pregnancy (if a women becomes pregnant during the study she will be excluded)
* Not being involve in sex work or being involved in sex work for more than 6 years
* Having a chronic disease
* Consumption of the medication listed in appendix entitled: list of other medication for health conditions
* Being allergic to acetylsalicylic acid, other medication for pain or fever, tartrazine or any other medication
* Having heartburn, stomach pain, stomach ulcer, anemia, hemophilia, kidney or liver disease, psoriasis, porphyria or other blood disease, G-6-PD deficiency, dermatitis (skin inflammation), alcoholism
* Having a history of a diagnosed cardiovascular event, heart failure, peripheral arterial disease, angina, stoke, transient ischemic attack
* Having a current or recurrent condition with a high risk of major bleeding
* Having anemia
* Current participation in a clinical trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Be a female. Having a female genital tract with a uterus
Enrollment: 300 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the proportion of HIV Target cells (CD4+CCR5+) | Baseline and at each month; For six months following enrolment
  Fresh cervical mononuclear cell populations from the cytobrush/scraper will be stained with monoclonal antibodies, and analyzed by flow cytometry. Proportion of CD4+CCR5+ T cells will be assessed at baseline and over the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Kenyan Aids Control Project/University of Nairobi, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No
we are not planing to share individuals data